CLINICAL TRIAL: NCT05689983
Title: Symptom-driven ICS/LABA Therapy for Adolescent Patients With Asthma Non-adherent to Daily Maintenance Inhalers
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202203033; KL2TR002346 (NIH); UL1TR002345 (NIH)
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children; Nonadherence, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomization will occur using a 1:1 ratio with random numbers generated using SAS 9.4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- As needed inhaled corticosteroid and long-acting beta-agonist (Active Comparator): Symptom-driven ICS/LABA treatment strategy
  Interventions: Drug: Symptom-driven budesonide/formoterol combination
- Standard therapy: maintenance inhaled corticosteroid and as needed short-acting beta-agonist (Placebo Comparator): Continue maintenance ICS and SABA therapy
  Interventions: Drug: Maintenance ICS and Symptom Driven SABA

INTERVENTIONS:
Drug: Maintenance ICS and Symptom Driven SABA — In this intervention, patients will be assigned to a standard therapy with a maintenance inhaled corticosteroid (Flovent) and an as needed short-acting beta-agonist and their adherence to this regimen will be assessed and compared to patients taking a regimen with an as needed inhaled corticosteroid and long-acting beta-agonist.
  Arms: Standard therapy: maintenance inhaled corticosteroid and as needed short-acting beta-agonist
Drug: Symptom-driven budesonide/formoterol combination — In this intervention, patients will be assigned to a symptom-driven budesonide/formoterol combination therapy (Symbicort) and their adherence to this regimen will be assessed and compared to patients taking a standard therapy with a maintenance inhaled corticosteroid and as needed short-acting beta-agonist.
  Arms: As needed inhaled corticosteroid and long-acting beta-agonist

SUMMARY:
Inhaler nonadherence is a common problem that has been estimated to account for approximately 60% of all asthma-related hospitalizations. Unfortunately, prior interventions to improve inhaler nonadherence have shown a lack of long-term success. This study proposes to assess the problem of non-adherence using a D&I research lens while testing a new inhaler approach to potentially ameliorate the detrimental consequences of maintenance inhaler nonadherence.

DETAILED DESCRIPTION:
While inhaled corticosteroids (ICS) are considered the essential foundation of most asthma therapy, ICS inhaler non-adherence is a notoriously common problem and a significant cause of asthma-related morbidity. Partially acknowledging the problem of non-adherence, international organizations recently made paradigm-shifting recommendations that all patients with mild or mild-to-moderate persistent asthma be considered for symptom-driven ICS-containing inhalers rather than relying on adherence to traditional maintenance ICS inhalers and symptom-driven beta-agonists. With this novel approach, asthma patients are at least exposed to the important anti-inflammatory effects of ICS-containing inhalers when their inhaler is deployed due to symptoms. The proposed study aims to (Aim 1) undertake a pragmatic pilot randomized-controlled trial to evaluate if an inhaler strategy that utilizes symptom-driven ICS inhalers is particularly accepted and beneficial in maintenance ICS inhaler non-adherent adolescent asthma patients, and (Aim 2) use a D&I science conceptual framework to better understand patients' and providers' views of inhaler non-adherence. This study will use an electronic sensor to monitor inhaler adherence and include semi-structured interviews using the Consolidated Framework for Implementation Research (CFIR).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide informed consent.
2. Age 18-75 at the time of study enrollment.
3. Provider diagnosed mild or moderate persistent asthma and prescribed maintenance ICS treatment and as needed SABA for at least 6 months prior to enrollment.
4. Suboptimal adherence to prescribed maintenance ICS therapy defined as missing at least expected 2 ICS refills in the prior 6 months based on examination of pharmacy records or a Medication Adherence Report Scale for Asthma (MARS-A) score <4.5.
5. An Asthma Control Test (ACT) score at enrollment greater than or equal to 12 but less than or equal to 20 indicating partially controlled or moderately uncontrolled asthma.
6. iPhone or Android smartphone with an active data plan and willingness to use the Adherium device.

Exclusion Criteria:

1. Relevant comorbid pulmonary diseases including, but not limited to a diagnosis of chronic obstructive pulmonary disease (COPD), cystic fibrosis, or alpha 1 anti-trypsin deficiency.
2. Current use of a biologic medication or investigational treatment for asthma.
3. History of asthma requiring ICU admission in the last year.
4. Unwillingness to use or pay for an inhaler that is compatible with the Adherium sensor (fluticasone propionate or budesonide/formoterol). Of note, fluticasone and budesonide/formoterol are formulary tier 1-2 for Missouri Medicaid and most commercial insurances and are believed to be equally or less expensive as alternative inhalers for most patients.
5. Any clinically significant abnormalities on physical exam, laboratory testing, or baseline diagnostic testing that the study team believes will make the study unsafe.
6. Patients who do not complete at least 70% of the twice-daily texts during the two weeks after screening.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to inhaler strategy delineated using an electronic inhaler sensor | 24 weeks
  The primary outcome will be adherence with an inhaler management strategy delineated using the Adherium inhaler sensor and smartphone application as compared between groups. Adherence to the treatment strategy for the maintenance ICS inhaler group will be calculated as the proportion of maintenance ICS actuations per prescription recommendation. Adherence for the symptom-based ICS treatment strategy will be calculated as the proportion of ICS/LABA actuations per recommendation based on self-report of symptoms (definition: ICS/LABA inhaler actuation during a day or night period divided by a period wherein a patient identified symptoms as >1 on REDCap-delivered smartphone questionnaire).

SECONDARY OUTCOMES:
Number of asthma exacerbations | 24 weeks
  Frequency of study-defined asthma exacerbations between groups (adjusted for time on treatment). Asthma exacerbations will be defined as an urgent medical visit for asthma symptoms, prescription of oral corticosteroids for asthma symptoms, or high use of a rescue inhaler (>16 actuations of SABA or >8 actuations of ICS/LABA within 24 hours on two consecutive days as assessed via the Adherium device).
Time to asthma exacerbation | 24 weeks
  Time to first exacerbation between groups. Asthma exacerbations will be defined as an urgent medical visit for asthma symptoms, prescription of oral corticosteroids for asthma symptoms, or high use of a rescue inhaler (>16 actuations of SABA or >8 actuations of ICS/LABA within 24 hours on two consecutive days as assessed via the Adherium device)
ICS exposure | 24 weeks
  Converted cumulative dose of ICS between groups.
Adverse and serious adverse events | 24 weeks
  Occurrence of any severe and non-severe adverse events between groups.
Change in Asthma Control Questionnaire (ACQ) | 24 weeks
  Change in Asthma Control Questionnaire (ACQ) from baseline to the final study visit. This is measured using the Asthma Control Questionnaire (ACQ) which is scaled from a minimum of 0 to a maximum of 6 for each question with higher scores indicating greater asthma control.
Change in asthma control test (ACT) | 24 weeks
  Change in Asthma Control Test (ACT) from baseline to the final study visit. This is measured using the Asthma Control Test (ACT) is scaled on a 5 point Likert scale from a minimum of 1 to a maximum of 5 for each question with higher scores indicating greater asthma control.
Change in Asthma Quality of Life Questionnaire (AQLQ) | 24 weeks
  Change in Asthma Quality of Life Questionnaire (AQLQ) from baseline to the final study visit. This is measured using the Asthma Quality of Life Questionnaire (AQLQ) which is scaled on a 7 point Likert scale from a minimum of 1 to a maximum of 7 for each question with higher scores indicating no impairment in activities due to asthma.
Change in Medication Adherence Reporting Scale for Asthma (MARS-A) questionnaire | 24 weeks
  Change in Medication Adherence Reporting Scale for Asthma (MARS-A) questionnaire from baseline to the final study visit. This is measured using the Medication Adherence Reporting Scale for Asthma (MARS-A) questionnaire which is scaled on a 5 point Likert scale from a minimum of 1 to a maximum of 5 for each question with higher scores indicating better adherence to medication.
Change in IQVIA Treatment Satisfaction Questionnaire for Medication (TSQM) | 24 weeks
  Change in IQVIA Treatment Satisfaction Questionnaire for Medication (TSQM) from baseline to the final study visit. This is measured using the IQVIA Treatment Satisfaction Questionnaire for Medication Version II (TSQM-2) which has 11 questions, 10 of which are scaled on a Likert scale from a minimum of 1 (Extremely Dissatisfied) to a maximum of 7 (Extremely Satisfied) with the exception of one question that asks about the experience of side effects in patients with answer choices of yes or no with higher scores indicating greater patient satisfaction with their medications.
Change in The Knowledge, Attitude, and Self-Efficacy Asthma Questionnaire (KASEAQ) | 24 weeks
  Change in The Knowledge, Attitude, and Self-Efficacy Asthma Questionnaire (KASEAQ) from baseline to the final study visit. This is measured using the Knowledge, Attitude, and Self-Efficacy Asthma Questionnaire (KASEAQ) which contains a series of statements in the domains of knowledge, attitude, and self-efficacy with answer choices of True, Mostly True, Sometimes True and Sometimes False, Mostly False, and False. Higher scores indicated greater knowledge of asthma and asthma management, greater optimism and willingness in self-management of asthma, and greater confidence in the ability to manage and control asthma.
Change in Feeling of Satisfaction with Inhaler (FSI-10) questionnaire | 24 weeks
  Change in Feeling of Satisfaction with Inhaler (FSI-10) questionnaire from baseline to the final study visit. This is measured using the Feeling of Satisfaction with Inhaler questionnaire (FSI-10) which contains 10 questions that are scaled on a 5 point Likert scale with answer options ranging from 1 (hardly at all) to 5 (very) with higher scores indicating greater satisfaction with the inhaler.

CONTACTS AND LOCATIONS:
Overall Officials: James Krings, MD MSc, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No